CLINICAL TRIAL: NCT02520063
Title: A Phase I/II Study of Preoperative (Neoadjuvant) Combination of Letrozole (Femara), Everolimus (Afinitor), and TRC105 in Postmenopausal Women With Newly Diagnosed Local or Locally Advanced Potentially Resectable Hormone-Receptor Positive and Her2 Negative Breast Cancer
Brief Title: Combination of Letrozole, Everolimus and TRC105 in Postmenopausal Women With Hormone-Receptor Positive and Her2 Negative Breast Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Novartis Pharmaceuticals (Industry); Tracon Pharmaceuticals Inc. (Industry)
Responsible Party: Principal Investigator, Christos Vaklavas, MD, Associate Professor, University of Utah
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: F150701004 (UAB 1514); UAB1514 (Other: University of Alabama at Birmingham (UAB))
Record Dates: First submitted 2015-07-30; First posted 2015-08-11 (Estimated); Results first posted 2023-08-21 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Breast Cancer
Keywords: hormone-receptor positive breast cancer; Her2 negative breast cancer; neoadjuvant; everolimus; TRC105; letrozole
MeSH Terms: conditions — Breast Neoplasms | interventions — Letrozole; Everolimus; carotuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Phase I Cohort 1 (Experimental): Letrozole 2.5 mg PO daily until surgery, everolimus 5 mg PO daily for 24 weeks, and TRC105 15 mg/kg IV q 2 weeks for 24 weeks
  Interventions: Drug: Letrozole; Drug: Everolimus; Drug: TRC105
- Phase I Cohort 2 (Experimental): Letrozole 2.5 mg PO daily until surgery, everolimus 10 mg PO daily for 24 weeks, and TRC105 15 mg/kg IV q 2 weeks for 24 weeks
  Interventions: Drug: Letrozole; Drug: Everolimus; Drug: TRC105
- Phase I Cohort -1 (Experimental): Letrozole 2.5 mg PO daily until surgery, everolimus 5 mg PO daily for 24 weeks, and TRC105 10 mg/kg IV q 2 weeks for 24 weeks
  Interventions: Drug: Letrozole; Drug: Everolimus; Drug: TRC105
- Phase II (Experimental): Letrozole 2.5 mg PO daily until surgery, everolimus 5 or 10 mg PO daily for 24 weeks, and TRC105 15 or 10 mg/kg IV q 2 weeks for 24 weeks. Dose and regimen to be determined based on data from the phase I component.
  Interventions: Drug: Letrozole; Drug: Everolimus; Drug: TRC105

INTERVENTIONS:
Drug: Letrozole — A dose of 2.5 mg of letrozole will be given orally once each day until one day before surgery. This drug is commercially available and is not provided by the study.
  Other Names: Femara
Drug: Everolimus — The dose of everolimus will be escalated from 5 mg to 10 mg daily depending upon the cohort in Phase I. It is administered as an oral pill to be taken once daily up until four weeks prior to surgery.
  Other Names: Afinitor
Drug: TRC105 — The dose for TRC105 is either 15 or 10 mg/kg to be given intravenously every two weeks and continued until four weeks prior to surgery.

SUMMARY:
This study will test how well a new combination of three drugs (Letrozole, Everolimus, and TRC105) is tolerated and how well it works in Stage 2 and 3 breast cancer when given prior to definitive surgery. Letrozole blocks the estrogen receptor expressed by many breast cancers while everolimus blocks signals that drive cancer cells to grow. TRC105 is an investigational drug that blocks the formation and growth of blood vessels that feed the cancer and promote its growth. The goal of this study is to investigate the safety and efficacy of this multitargeted approach in breast cancer.

DETAILED DESCRIPTION:
In postmenopausal women with hormone receptor-positive and Her2 negative non-metastatic breast cancer, downstaging or the achievement of a complete pathologic remission before definitive surgery has been associated with the lowest risk of recurrence of breast cancer. In order to achieve a better response in these patients in the preoperative setting, this study combines 3 potentially synergistic agents. Letrozole blocks the synthesis of estrogens and, in doing so, deprives the tumor from hormones which drive its growth. Everolimus is a drug that blocks growth factor signaling which is essential for tumor cells to maintain their growth and proliferation. Everolimus has already been shown to work very well in this subtype of breast cancer in the recurrent and metastatic setting. TRC105 is an investigational agent that prevents the formation and growth of new blood vessels that support tumors by providing oxygen and nutrients.

The study has 2 components. First the investigators will determine the ideal in terms of tolerance combination of doses of the 3 agents. Once the ideal regimen is determined, more patients will be treated with the investigational combination. During this second stage, the investigators will get a preliminary idea of how effective the investigational therapy is. Further studies will need to be done to confirm the efficacy of the investigational combination.

ELIGIBILITY:
Inclusion Criteria:

* Recent diagnosis of hormone receptor positive and HER2 negative breast cancer.
* Stage 2 and 3 hormone receptor positive and HER2 negative breast cancer (stage T2-4 but not inflammatory, N0-2, M0).
* Histological grade I, II or III according to the modified Bloom Richardson scale.
* No prior treatment specific for breast cancer.
* Postmenopausal status as defined by the National Comprehensive Cancer Network.
* ECOG performance status < 2 (Karnofsky > 60%).
* Must have signed study-specific informed consent.
* Liver Function Tests < 2.5 times the upper normal limit (UNL).
* ANC ≥ 1,500/mm3, platelets ≥ 100,000/mm3, Hemoglobin ≥ 10g%.
* Renal function: serum creatinine < 1.5 institutional UNL or creatinine clearance > 40 cc/min.

Exclusion Criteria:

* Inflammatory breast cancer.
* Pre- and peri-menopausal state.
* Pregnancy.
* Metastatic disease.
* HER2 positive breast cancer by immunohistochemistry or FISH.
* Triple negative breast cancer (hormone receptor and Her2 negative).
* Disease that cannot be followed by imaging studies.

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-02-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erica Stringer-Reasor, M.D., Principal Investigator — University of Alabama at Birmingham; Erica Stringer-Reasor, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Vaklavas C, Stringer-Reasor EM, Elkhanany AM, Ryan KJ, Li Y, Theuer CP, Acosta EP, Wei S, Yang ES, Grizzle WE, Forero-Torres A. A phase I/II study of preoperative letrozole, everolimus, and carotuximab in stage 2 and 3 hormone receptor-positive and Her2-negative breast cancer. Breast Cancer Res Treat. 2023 Apr;198(2):217-229. doi: 10.1007/s10549-023-06864-9. Epub 2023 Feb 3. PMID 36735117

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase I Cohort 1: Letrozole: 2.5 mg was given orally once each day until one day before surgery. Everolimus: 5 mg was administered as an oral pill once daily until four weeks prior to surgery (24 weeks).
  TRC105: 15 mg/kg was given intravenously every two weeks and continued until four weeks prior to surgery (24 weeks).
- Phase I Cohort 2; Phase II: Letrozole: 2.5 mg was given orally once each day until one day before surgery. Everolimus: 10 mg was administered as an oral pill once daily until four weeks prior to surgery (24 weeks).
  TRC105: 15 mg/kg was given intravenously every two weeks and continued until four weeks prior to surgery (24 weeks).
- Phase I Cohort -1: Letrozole: 2.5 mg was given orally once each day until one day before surgery. Everolimus: 5 mg was administered as an oral pill once daily until four weeks prior to surgery (24 weeks).
  TRC105: 10 mg/kg was given intravenously every two weeks and continued until four weeks prior to surgery (24 weeks).
Period: Overall Study
Arm/Group | Phase I Cohort 1 | Phase I Cohort 2 | Phase I Cohort -1 | Phase II
Started | 6 | 4 | 0 | 5
Completed | 5 | 3 | 0 | 5
Not Completed | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Phase 1 Cohort -1 had no patients enrolled. as there was not enough toxicities to warrant a dose reduction.
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase I Cohort 1 | Phase I Cohort 2 | Phase I Cohort -1 | Phase II | Total
Number analyzed (Participants) | 6 | 4 | 0 | 5 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 4 | 0 | 3 | 13
  >=65 years | 0 | 0 | 0 | 2 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 0 | 5 | 15
  Male | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 5 | 4 | 0 | 4 | 13
  Black | 1 | 1 | 0 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced Dose-limiting Toxicities
Description: This outcome will report the number of patients who experienced a dose-limiting Toxicity (DLT) in Phase I Cohort 1, Phase I Cohort 2, and Phase I Cohort -1. A DLT was defined as:
  1. A grade 3 or 4 non-hematologic toxicity except anorexia, alopecia, nausea (which is not refractory to antiemetics), fatigue, and fever without neutropenia;
  2. Failure to recover to baseline (except alopecia) after delaying the next dose by more than 14 days;
  3. Grade 3 or 4 neutropenia complicated by fever >38.5°C or infection, or grade 4 neutropenia of ≥7 days duration; or
  4. Grade 4 thrombocytopenia, or grade 3 thrombocytopenia complicated by hemorrhage.
  The maximum tolerated dose (MTD) is defined as the highest dose at which 0 out of the first 3 or 1 out of a total of 6 patients experience DLT during the first cycle of therapy; this dose level will be the recommended phase 2 dose (RP2D) in the Phase II Group.
Time Frame: 4 weeks
Population: There were no patients enrolled in the phase 1 cohort -1 portion of the protocol due to lack of toxicities in phase 1 cohort 1 and 2.
Measure: Number; unit: participants
Arm/Group | Phase I Cohort 2 | Phase I Cohort 1 | Phase I Cohort -1
Number analyzed (Participants) | 4 | 6 | 0
participants | 0 | 1 |
Statistical Analysis 1: Comparison: Phase I Cohort 2 vs Phase I Cohort 1; Test type: Other; The primary analysis was of safety and included all patients who received at least one dose of the investigational regimen. The rate of adverse events was be estimated at the end of the study along with two-sided 95% exact CIs (Clopper-Pearson intervals)

2. Secondary Outcome: Rates of Pathologic Complete Remission (pCR)
Description: The 2-dimensional size of the surgically excised residual tumor was measured and compared to the radiographic size of the tumor at baseline.
  Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI:
  Complete Response (CR), Disappearance of all target lesions and reduction in short axis of any pathological lymph nodes to <10 mm; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: 24 weeks up to time of surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I Cohort 1 | Phase I Cohort 2 | Phase II
Number analyzed (Participants) | 6 | 4 | 5
Participants | 0 | 0 | 0

3. Secondary Outcome: C Max - Letrozole
Description: Maximum serum concentration of Letrozole.
Time Frame: Day 1 and Day 29
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/ml
Arm/Group | Phase I Cohort 1 | Phase I Cohort 2 | Phase II
Number analyzed (Participants) | 6 | 4 | 5
ng/ml
  Day 1 | 45.3 (31.5) | 41.2 (28.6) | 33.3 (43.8)
  Day 29 | 211 (32.7) | 292 (53.1) | 168 (73.5)

4. Secondary Outcome: Tumor Proliferation Changes
Description: This outcome will report the change in tumor cell proliferation. This was measured by the change in the percentage of Ki67 positive cells from pretreatment to surgery (up to 24 weeks): (%Ki67(+) cells pretreatment - %Ki67(+) cells posttreatment)/(%Ki67(+) cells pretreatment) * 100 Ki67 is a protein found in cells that are dividing. The Ki-67 assessment was performed by the clinical histology laboratory using a validated assay. The results were evaluated by a board-certified pathologist, who estimated the proportion of cancer cells stained for Ki-67. The individual tissue sections were analyzed blindly and at the completion of the assay, results were correlated per case as to changes in Ki-67 with the investigational therapy.
Time Frame: 24 weeks (pretreatment to time of definitive surgery)
Population: There were no patients enrolled in Phase 1 Cohort -1 due to the lack of toxicities in Phase 1 Cohort 1 and Phase I Cohort 2. Additionally, one patient in Phase 1 Cohort 1, one patient in Phase 1 cohort 2, and two patients in Phase 2 were not evaluable for this outcome measure.
Measure: Median (Full Range); unit: percent change in the of Ki67(+) cells
Arm/Group | Phase I Cohort 1 | Phase I Cohort 2 | Phase II
Number analyzed (Participants) | 5 | 3 | 3
percent change in the of Ki67(+) cells | -96.7 [-100 to -83.3] | 14 [-100 to 240] | -77.8 [-100 to -38.5]

5. Secondary Outcome: T Max - Letrozole
Description: T Max is the time to the maximum serum concentration of a drug in the blood. This outcome will report the T Max of Letrozole at Day 1 in Phase 1 Cohort 1, Phase 1 Cohort 2, and Phase 2. All patients in the trial received the same dose of letrozole.
Time Frame: Day 1
Measure: Median (Full Range); unit: Hours
Groups:
- Phase 2: Letrozole: 2.5 mg was given orally once each day until one day before surgery. Everolimus: 10 mg was administered as an oral pill once daily until four weeks prior to surgery (24 weeks).
  TRC105: 15 mg/kg was given intravenously every two weeks and continued until four weeks prior to surgery (24 weeks).
Arm/Group | Phase I Cohort 1 | Phase I Cohort 2 | Phase 2
Number analyzed (Participants) | 6 | 4 | 5
Hours | 3 [2 to 24] | 1.5 [1 to 2] | 2 [1 to 4]

6. Secondary Outcome: AUC - Letrozole
Description: This outcome will report the area under the serum concentration of letrozole versus time curve (AUC-L).
  AUC-L is the integral of the concentration of letrozole in the blood as a function of time. AUC-L measures how much letrozole reaches the bloodstream in a period of time after a dose is given. This is useful in dose determination and assessing drug interactions.
  This outcome was assessed on Day 1 and on Day 29 for Phase I Cohort I, Phase I Cohort 2, and Phase 2.
Time Frame: Day 1 and Day 29
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hrs/ml
Arm/Group | Phase I Cohort 1 | Phase I Cohort 2 | Phase 2
Number analyzed (Participants) | 6 | 4 | 5
ng*hrs/ml
  Day 1 | 639 (34) | 532 (17.1) | 408 (28.5)
  Day 29 | 3500 (41.7) | 2500 (205) | 1400 (195)

7. Secondary Outcome: T 1/2 - Letrozole
Description: T ½ is the half-life of a drug in the blood. This is the time it takes for the concentration of the drug in the blood to be reduced by half. This outcome will report the T 1/2 of Letrozole.
Time Frame: Day 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Phase I Cohort 1 | Phase I Cohort 2 | Phase 2
Number analyzed (Participants) | 6 | 4 | 5
Hours | 15.5 (4.26) | 24.7 (2.34) | 31.7 (11.4)

8. Secondary Outcome: C Max - Everolimus
Description: Cmax is the maximum serum concentration of a drug in the blood. This outcome will report the Cmax of Everolimus in Phase 1 Cohort 1 and Phase 1 Cohort 2 combined with Phase 2 (since the dose of everolimus was the same in these cohorts) at Day 1 and Day 29.
Time Frame: Day 1 and Day 29
Population: Phase 1 Cohort 1 and Phase 1 Cohort 2 combined with Phase 2 (since the dose of everolimus was the same in these cohorts) at Day 1 and Day 29.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Phase I Cohort 2 and Phase 2: Letrozole: 2.5 mg was given orally once each day until one day before surgery. Everolimus: 10 mg was administered as an oral pill once daily until four weeks prior to surgery (24 weeks).
  TRC105: 15 mg/kg was given intravenously every two weeks and continued until four weeks prior to surgery (24 weeks).
Arm/Group | Phase I Cohort 1 | Phase I Cohort 2 and Phase 2
Number analyzed (Participants) | 6 | 9
ng/mL
  day 1 | 1.56 (51.5) | 3.7 (55.5)
  day 29 | 2.63 (27.9) | 5.38 (86.7)

9. Secondary Outcome: T Max Everolimus
Description: T Max is the time to the maximum serum concentration of a drug in the blood. This outcome will report the T Max of Everolimus in Phase 1 Cohort 1, and combined Phase 1 Cohort 2 and Phase 2 (since patients received the same dose of everolimus) at Day 1.
Time Frame: Day 1
Population: Phase 1 Cohort 1, and combined Phase 1 Cohort 2 and Phase 2 (since patients received the same dose of everolimus) at Day 1
Measure: Median (Full Range); unit: hours
Arm/Group | Phase I Cohort 1 | Phase I Cohort 2 and Phase 2
Number analyzed (Participants) | 6 | 9
hours | 2 [1 to 6] | 1 [1 to 4]

10. Secondary Outcome: AUC - Everolimus
Description: This outcome will report the area under the serum concentration everolimus of versus the time curve (AUC-E).
  AUC-E is the integral of the concentration of everolimus in the blood as a function of time. AUC-E measures how much everolimus reaches the bloodstream in a period of time after a dose is given. This is useful in dose determination and assessing drug interactions.
  This outcome was assessed on Day 1 and on Day 29 for Phase I Cohort I, and combined Phase I Cohort 2 and Phase 2 (since patients in Phase I cohort 2 and Phase 2 received the same dose of everolimus).
Time Frame: Day 1 and Day 29
Population: Phase I Cohort I, and combined Phase I Cohort 2 and Phase 2 (since patients in Phase I cohort 2 and Phase 2 received the same dose of everolimus)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hrs/mL
Arm/Group | Phase I Cohort 1 | Phase I Cohort 2 and Phase 2
Number analyzed (Participants) | 6 | 9
ng*hrs/mL
  Day 1 | 15.4 (41.9) | 20.9 (50.4)
  Day 29 | 22.5 (39.3) | 32.1 (153)

11. Secondary Outcome: T 1/2 - Everolimus
Description: T ½ is the half-life of a drug in the blood. This is the time it takes for the concentration of the drug in the blood to be reduced by half. This outcome will report the T 1/2 of Everolimus in Phase 1 Cohort 1 and combined Phase 1 Cohort 2 and Phase 2 at Day 1 (since patients in Phase 1 Cohort 2 and Phase 2 at Day 1 received the same dose of everolimus).
Time Frame: day 1
Population: Phase 1 Cohort 1 and combined Phase 1 Cohort 2 and Phase 2 at Day 1 (since patients in Phase 1 Cohort 2 and Phase 2 at Day 1 received the same dose of everolimus).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Phase I Cohort 1 | Phase I Cohort 2 and Phase 2
Number analyzed (Participants) | 6 | 9
hours | 13.4 (1.64) | 11.8 (7.86)

ADVERSE EVENTS:
Time Frame: 6 months
Description: There were no patients enrolled in the phase 1 cohort -1 section due to lack of adverse events in phase 1 cohorts 1 and 2.
Arm/Group | Phase I Cohort 1 | Phase I Cohort 2 | Phase I Cohort -1 | Phase II
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/4 | 0/0 | 0/5
Serious Adverse Events (participants affected / at risk) | 1/6 | 0/4 | 0/0 | 0/5
Other Adverse Events (participants affected / at risk) | 6/6 | 4/4 | 0/0 | 0/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I Cohort 1 (N=6) | Phase I Cohort 2 (N=4) | Phase I Cohort -1 (N=0) | Phase II (N=5)
headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I Cohort 1 (N=6) | Phase I Cohort 2 (N=4) | Phase I Cohort -1 (N=0) | Phase II (N=5)
headache (Nervous system disorders) | 6 (6) | 4 (4) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-07-25): https://cdn.clinicaltrials.gov/large-docs/63/NCT02520063/Prot_SAP_002.pdf
  • Informed Consent Form (2019-07-25): https://cdn.clinicaltrials.gov/large-docs/63/NCT02520063/ICF_003.pdf